CLINICAL TRIAL: NCT02894645
Title: Ma-Spore ALL 2010 Study
Brief Title: Malaysia-Singapore Acute Lymphoblastic Leukemia 2010 Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ma-Spore ALL 2010
Record Dates: First submitted 2016-08-25; First posted 2016-09-09 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Acute Lymphoblastic Leukemia (ALL)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Prednisolone; Dexamethasone; Asparaginase; Vincristine; Methotrexate; Daunorubicin; Doxorubicin; Cyclophosphamide; Cytarabine; Mercaptopurine; Thioguanine; fludarabine; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Risk (SR) (Other)
  Interventions: Drug: Prednisolone; Drug: Dexamethasone; Drug: L-Asparaginase; Drug: Vincristine; Drug: Methotrexate; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: 6-Mercaptopurine; Drug: Thioguanine
- Intermediate Risk (IR) (Other)
  Interventions: Drug: Prednisolone; Drug: Dexamethasone; Drug: L-Asparaginase; Drug: Vincristine; Drug: Methotrexate; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: 6-Mercaptopurine; Drug: Thioguanine
- High risk (HR) (Other)
  Interventions: Drug: Prednisolone; Drug: Dexamethasone; Drug: L-Asparaginase; Drug: Vincristine; Drug: Methotrexate; Drug: Daunorubicin; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: 6-Mercaptopurine; Drug: Thioguanine; Drug: Fludarabine; Drug: Imatinib

INTERVENTIONS:
Drug: Prednisolone — Oral
Drug: Dexamethasone — Oral
Drug: L-Asparaginase — Intramuscular injection
Drug: Vincristine — Intravenous
Drug: Methotrexate — Intrathecal/ Intravenous/ Oral
Drug: Daunorubicin — Intravenous
  Arms: High risk (HR)
Drug: Doxorubicin — Intravenous
  Arms: High risk (HR); Intermediate Risk (IR)
Drug: Cyclophosphamide — Intravenous
Drug: Cytarabine — Intravenous/ Subcutaneous injection
Drug: 6-Mercaptopurine — Oral
Drug: Thioguanine — Oral
Drug: Fludarabine — Intravenous
  Arms: High risk (HR)
Drug: Imatinib — Oral (For BCR-ABL ALL only)
  Arms: High risk (HR)

SUMMARY:
The overall objective of this study is to continue to improve the cure rate of childhood acute lymphoblastic leukemia (ALL) in Singapore and Malaysia in the context of a multi-centre cooperative trial using a risk-stratified therapy based primarily on early response to therapy utilizing a simplified minimal residual disease (MRD-lite) platform.

DETAILED DESCRIPTION:
The study was designed on the premise that a risk classification strategy combining clinical and genetic presenting features with molecular assessment of MRD should reduce both treatment-related toxicities and relapse risk.

The patient will be assigned to one of the 3 risk groups depending on his/her response to the treatment and special laboratory tests. There are no experimental drugs in this study. All the drugs used are standard established treatment for childhood ALL for the last 30 years. The difference in treatment is by changes in the frequency and dose of the chemotherapy drugs.

The overall study treatment lasts for about 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of non-Burkitt B-lineage ALL
2. 1 to 17 years of age (before 18th birthday)
3. Renal function within normal range for age
4. Liver function within normal range for age
5. Able to participate in the full 2 years of treatment

Exclusion Criteria:

1. Age less than one year or age greater than/equals to 18 years
2. Previous treatment with cytotoxic agents or high-dose steroids
3. Mixed phenotype acute leukemia (MPAL)
4. ALL as secondary malignancy
5. Abnormal renal or liver function
6. Doubtful compliance or unable to afford full course of therapy

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2008-10; Primary Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 5 years
  EFS was estimated from time of diagnosis to time of first event or of patient's last follow-up. Failure to achieve complete remission (CR), relapse, death in continuous remission from whatever cause, secondary leukemia and abandonment (absence from scheduled therapy for more than 6 weeks) were considered as events.
Overall survival (OS) | 5 years
  OS was determined from diagnosis to time of death from any cause.
Minimal residual disease (MRD) measurement | At time point of Day 33, week 8 and week 12

SECONDARY OUTCOMES:
Number of participants with chemotherapy-related adverse events as assessed by CTCAE version 4.0 | Through study completion, an average of 2 years
Dose intensity of chemotherapy during various phases of therapy | Through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Allen Yeoh, MBBS, Principal Investigator — Ma-spore Group
Locations (4):
- Malaysia (2):
  - University of Malaya Medical Centre, Kuala Lumpur
  - Subang Jaya Medical Centre, Subang Jaya
- Singapore (2):
  - National University Hospital, Singapore
  - KK Women's and Children's Hospital, Singapore

REFERENCES:
- [Derived] Ariffin H, Chiew EKH, Oh BLZ, Lee SHR, Lim EH, Kham SKY, Abdullah WA, Chan LL, Foo KM, Lam JCM, Chan YH, Lin HP, Quah TC, Tan AM, Yeoh AEJ. Anthracycline-Free Protocol for Favorable-Risk Childhood ALL: A Noninferiority Comparison Between Malaysia-Singapore ALL 2003 and ALL 2010 Studies. J Clin Oncol. 2023 Jul 10;41(20):3642-3651. doi: 10.1200/JCO.22.02347. Epub 2023 Jun 5. PMID 37276496
- [Derived] Yeoh AEJ, Lu Y, Chin WHN, Chiew EKH, Lim EH, Li Z, Kham SKY, Chan YH, Abdullah WA, Lin HP, Chan LL, Lam JCM, Tan PL, Quah TC, Tan AM, Ariffin H. Intensifying Treatment of Childhood B-Lymphoblastic Leukemia With IKZF1 Deletion Reduces Relapse and Improves Overall Survival: Results of Malaysia-Singapore ALL 2010 Study. J Clin Oncol. 2018 Sep 10;36(26):2726-2735. doi: 10.1200/JCO.2018.78.3050. Epub 2018 Jul 25. PMID 30044693